CLINICAL TRIAL: NCT05405933
Title: Comparison of Propioceptive Neuromuscular Facilitation Vs Balance Exercise Along With Conventional Therapy for Balance and Gait in Chronic Parkinson's Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/512
Record Dates: First submitted 2022-05-09; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Parkinson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propioceptive Neuromuscular Facilitation (Experimental): Propioceptive Neuromuscular Facilitation With Conventional Therapy for Balance and Gait
  Interventions: Diagnostic Test: Propioceptive Neuromuscular Facilitation
- Balance Exercise (Experimental): Balance Exercise Along With Conventional Therapy for Balance and Gait
  Interventions: Diagnostic Test: Balance Exercise

INTERVENTIONS:
Diagnostic Test: Propioceptive Neuromuscular Facilitation — Propioceptive Neuromuscular Facilitation With Conventional Therapy for Balance and Gait
  Arms: Propioceptive Neuromuscular Facilitation
Diagnostic Test: Balance Exercise — Balance Exercise Along With Conventional Therapy for Balance and Gait
  Arms: Balance Exercise

SUMMARY:
To determine the effect of Proprioceptive Neuromuscular Facilitation Vs Balance Exercise along with Conventional Therapy for balance and gait in Chronic Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Parkinson's patients.(34)
* Patients from both gender around the age of 45-65.(35)
* Patient with a score of 42 above on the Berg Balance Scale.(29)
* Patient with good cognitive function minimum score of 20 or more on Mini-mental Status Examination Scale (MMSE).(36)

Exclusion Criteria:

* Patients with a history of recurrent stroke.(37)
* Patient with peripheral vascular disease.(38)
* Patient with fracture or dislocation of lower limb.(39)
* Patient with peripheral nerve injury.(40)
* Patient with skin discoloration, skin ulcers, and skin allergy.(41)

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Balance Exercise Along With Conventional Therapy | 6 Months
  30 participants in Balance Exercise with routine Physical therapy for 45 minutes on lower limb. The interventions will be performed by a trained physiotherapist. Berg Balance Scale, Functional Gait Assessment Tool
Propioceptive Neuromuscular Facilitation | 6 Months
  30 participants in Proprioceptive Neuromuscular Facilitation with routine Physical Therapy for 45 minutes on lower limb. Minimental Status Examination Tool.

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital Jinnah hospital Mayo hospital Chaudhry Muhammad Akram Teaching and research hospital Services hospital Lahore (SHL), Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No